CLINICAL TRIAL: NCT03464747
Title: Continuous Central Venous Lactate Monitoring by Intravascular Microdialysis : a Comparison to Sequential Arterial Lactate Measurement During Shock.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB : 16.09.02
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Shock
Keywords: Lactic Acid
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EIRUS system (Maquet Critical Care AB, 17154, Solna, Sweden) — continuous measurement of venous lactate through a central venous catheter by microdialysis

SUMMARY:
During shock, arterial hypotension, inadequate cardiac output and microcirculatory alterations lead to tissue hypoxia, multiple organ failure and death. Arterial lactate is considered as the best marker of tissue hypoxia. A lactate decrease during the first 6 hour is strongly associated with better outcome and may be used as a target for assessing the efficiency of shock resuscitation.

The EIRUS system (Maquet Critical Care AB, 17154, Solna, Sweden) is a new device allowing the continuous measurement of venous lactate through a central venous catheter.

However, before being used extensively, such device needs to be evaluated concerning its accuracy. The aim of the present study is to assess the reliability of this device.

ELIGIBILITY:
Inclusion Criteria:

Acute circulatory failure defined as : systolic blood pressure<90mmHg or mean arterial pressure <65mmHg and blood lactate > 2mmol/L

Exclusion Criteria: Pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Agreement | Every 4hours for 48hours
  Agreement between sequential arterial blood lactate measurement and continuous venous lactate obtained by microdialysis

SECONDARY OUTCOMES:
Interchangeability | Every 4hours for 48hours
  Interchangeability of the variations of the two methods using the trend interchangeability method

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: Undecided